CLINICAL TRIAL: NCT02850393
Title: Etude en Imagerie Par résonance magnétique Fonctionnelle et Structurelle Des mécanismes de Suppression mnésique Dans Les Troubles Obsessionnels Compulsifs
Brief Title: Inhibitory Control of the Mind : Neural Bases and Impact for Obsessive-compulsive Disorders
Acronym: SUPTOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre National de la Recherche Scientifique, France (Other); Université de Caen Normandie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-A01609-40; 160028B-31 (Other: ANSM)
Record Dates: First submitted 2016-05-27; First posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Obsessive Compulsive Disorder; Healthy
Keywords: suppression mnemonic; emotional response; inhibitory control of failures; neurological alterations
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patients with obsessive compulsive disorder (Experimental): Functional magnetic resonance imaging behavioral measures physiological measurements
  Interventions: Other: Functional magnetic resonance imaging; Behavioral: behavioral measures; Other: physiological measurements
- healthy participants (Experimental): Functional magnetic resonance imaging behavioral measures physiological measurements
  Interventions: Other: Functional magnetic resonance imaging; Behavioral: behavioral measures; Other: physiological measurements

INTERVENTIONS:
Other: Functional magnetic resonance imaging
Behavioral: behavioral measures
Other: physiological measurements

SUMMARY:
Mental-health conditions affect million people worldwide. The economic burden of mental illness is enormous and the economic health of both developing and developed nations will depend on controlling the staggering growth in costs from mental disorders. Obsessive-compulsive disorder (OCD) is a relatively common and frequent form of anxiety that affects approximately 2-3% of the population. OCD is characterized by anxiety, obsessions (persistent intrusive thoughts and images with highly distressing contents) and compulsions (repetitive activity), and severely impairs the lives of those affected. Despite their interest as effective and affordable care and rehabilitation, cognitive therapeutic profits too little from the increasing accumulation of knowledge in neuroscience, and neuroscientists pay too little attention to the challenges faced by clinical psychologists and psychiatrists. To reduce this cultural gap, two teams specialized in the study and multimodal imaging of healthy participants and clinical patients with mental health disorders, the UMR-S INSERM-EPHE-UNICAEN U1077 unit led by Francis Eustache, and ISTS team (UMR-S 6301 CNRS-CEA-UCBN) led by Sonia Dollfus, will joint their efforts to develop an integrated approach of the neural mechanisms at stake from basic neuroscience using state-of-art neuroimaging techniques, to novel and ground breaking psychological intervention. Both teams evolve at the brain imaging Cyceron center in Caen in connection with the Mental Health and Addictology Center, offering unique opportunities for such translational research. This project will capitalize on recent evidence showing that healthy participants can prevent unwanted images from entering consciousness using inhibitory control and memory suppression techniques, disrupting traces of the memories in sensory areas of the brain, and weakening their vividness and later reentrance. OCD is characterized by aberrant and excessive visual intrusions, usually extremely vivid, detailed, and unpleasant. These distressing images are particularly uncontrollable and may frequently initiate compulsive rituals. In a first phase of this proposal will use functional magnetic resonance imaging (fMRI) to develop a neurobiological model of the cognitive computations achieved by inhibition network to suppress memory. To achieve this goal we will develop an attentional model of healthy memory inhibition functioning, simulating the deployment of attentional resources and the different mental processes at stake during suppression. Using sophisticated analyzing tools of fMRI data, we will use this model to decode and infer the representational content of the brain inhibition network, and further refine the connectivity pathways which underlie such control. The lack of a strong neurobiological model prevents the development of therapies which would increase functionality of this network and optimize intervention aiming to disrupt mental intrusions and obsessions. In a second phase, we will assess whether memory suppression may be transferred and trained in OCD patients using images depicting their own obsessions, as a promising avenue to reduce their symptoms on the long run. In addition, fMRI and other brain structural acquisitions will be collected before and after cognitive training to memory suppression, offering a unique opportunity to observe the online dysfunction of intrusion control in OCD patients and to identify neurobiological markers predictive of training outcome and network reconfiguration with training. A fundamental goal of motivated forgetting involves not only to exclude unwelcome content from consciousness but also to reduce their later emotional impact by doing so. In parallel of these two main phases, we will thus also measure physiological markers of autonomic nervous system activity changes in response to suppressed images to better identify the consequences of memory suppression on emotional states, anxiety, and mental health in general.

ELIGIBILITY:
Inclusion Criteria :

* All the participants :

  * Participants between 18 and 55 years old
  * Affiliated to the French national health care system
  * French native speaker
  * Right-handed
  * At least education after graduating with french GSCE "brevet des collèges"
  * Body mass < 35kg/m2
* Healthy subjects :

  * Signed written consent form
* Patients :

  * Patients with OCD according to DSM V diagnostic criteria at the time of the study
  * Stabilized (no change of psychotropic drugs during the last 3 months)
  * Signed written consent form associated with the agreement of the tutor and / or curator for protected adults

Exclusion Criteria:

* All the participants :

  * Pregnancy or intent to get pregnant
  * Person deprived of their liberty
  * Person admitted to a health or social institution for purposes other than research
  * Minor
  * Protected adults or people unable to give informed consent
  * Person subjected to an exclusion period related to another protocol
  * History of cancer with the last 5 years, excluding squamous cell carcinomas
  * Alcoholism, antecedents of chronic alcoholism or drugs abuse
  * Use of medication that may interfere with cognitive or cerebral functioning
  * Presence of visual or hearing troubles that may compromise participant's ability to participate in the study
  * MRI Contraindications
* Healthy subjects :

  * History of neurological or psychiatric disorders or existence of traumatic brain injury with loss of consciousness for more than one hour
  * Severe psychiatric disorders (according to DSM V diagnostic criteria) or psychological troubles which could affect participant's judgment
* Patients :

  * Presence of neurological history, history of head trauma with loss of consciousness for more than an hour, severe depression, manic symptoms, post-traumatic stress, borderline personality disorder, antisocial, paranoid or schizoid.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-03 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Blood Oxigen Level Dependent (BOLD) response as measured with fMRI | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Anaïs Vandevelde, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- GIP Cyceron, Caen, Calvados, France